CLINICAL TRIAL: NCT02325089
Title: Effect of Treating Sleep Apnea With Oral Appliances in the Elderly: ORACLE Study
Brief Title: ORal ApplianCes for sLeep Apnea of the Elderly
Acronym: ORACLE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Denis Martinez, MD, PhD, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 140069
Record Dates: First submitted 2014-10-28; First posted 2014-12-24 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Obstructive Sleep Apnea; Hypertension; Cardiovascular Disease
Keywords: Elderly; Obstructive Sleep Apnea; Mandibular advancement oral appliance; Hypertension; Cardiovascular disease; Quality of life
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension; Cardiovascular Diseases | interventions — Occlusal Splints

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mandibular advancement device (Experimental): Mandibular advancement device titrated to reduce or eliminate snoring and sleep apnea
  Interventions: Device: Mandibular advancement device
- Placebo (Placebo Comparator): Oral appliance identical to the mandibular advancement device without mandibular advancement
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Mandibular advancement device — Use of a mandibular advancement device every night during one year. Device will be titrated to reduce or - if possible - eliminate snoring and sleep apnea.
  Other Names: MAD
  Arms: Mandibular advancement device
Device: Placebo — Placebo oral appliance will be identical to the mandibular advancement device without, however, the attachemnt to allow mandibular advancement. It will be used every night during one year.
  Other Names: Placebo device
  Arms: Placebo

SUMMARY:
Sleep apnea involves significant increases in disease and death, but its consequences in people over 65 years of age are incompletely recognized. Intraoral mandibular advancement appliances reduce the number of apneas and hypopneas. The investigators hypothesized that oral appliances provided to the elderly may prevent hypertension and other consequences of sleep apnea in large populations, at a favorable cost/benefit relationship for the public health system.

DETAILED DESCRIPTION:
Sleep disorders involve significant increases in morbidity and mortality, particularly in those over 60 years. Sleep apnea is the leading identifiable cause of hypertension, which is the main cause of cardiovascular disease. Some degree of sleep apnea is present in up to 95% of the elderly. Intraoral mandibular advancement appliances reduce the number of apneas and hypopneas.

We hypothesized that reducing the number of sleep apnea events through oral appliances is effective in preventing high blood pressure and other consequences of sleep apnea in the elderly in the public health system setting. In this superiority parallel, randomized, and double-blinded study we will compare the effect of an intraoral appliance with mandibular advancement to a placebo device without mandibular advancement in preventing high blood pressure and other consequences of sleep apnea in the elderly. The duration of intervention will be of 12 months, with assessments at three, six months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Mandibular advancement of at least 3 mm
* Mouth opening of at least 30 mm
* Sleep apnea with apnea-hypopnea index between 10 and 50 events/hour
* Agree to participate in the study by signing the informed consent

Exclusion Criteria:

* Already in treatment for sleep apnea
* Self-reported severe or terminal Illness
* Physical disability
* Inability to communicate verbally
* Dementia in the Mini-Mental State Examination
* Plan to move to a different a city or to be institutionalized in the next year
* Participation in another clinical trial
* Less than eight teeth, periodontal disease, or TMJ problems

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Arterial Blood Pressure Monitoring (ABPM) | 12 months
  24-h, diurnal, and sleep systolic and diastolic blood pressure. Systolic and diastolic dipping.

SECONDARY OUTCOMES:
Composite measure of Metabolic Syndrome including Glucose, Cholesterol, Triglyceride, Blood pressure, and Waist circumference | 12 months
  The NCEP ATP III panel defined metabolic syndrome as the presence of three or more of the following risk determinants:
  1) triglyceride levels > to 150 mg / dl; 2) HDL-cholesterol < 40 for men and < 50 for women; 3) glucose > to 110 mg / dl; 4) blood pressure: Systolic > 130 mmHg and / or diastolic blood pressure > 85 mm Hg; 5) waist circumference > 88 cm in women and > 102 cm in men.
Composite measure of Physical Ability | 12 months
  The following areas will be evaluated: 1) functional capacity (six-minute walk test), 2) balance (Berg balance scale: 14-item scale designed to measure balance of the older adult in a clinical setting.), 3) flexibility (Wells Sit and Reach Test), 4) mobility (timed up and go test), 5) Force-Velocity Characteristics of Upper and Lower Limbs (Handgrip strength testing: upper, and Sit-to-stand test: Lower), 6) Recall of falls in the last six months
Composite measure of Pain | 12 months
  The pain assessment will be conducted by the following methods: 1) Profile of Chronic Pain 2) Assessment of Pain Catastrophizing
Quality of life measured by WHOQOL | 12 months
  The patients will answer the WHOQOL-Old module with 24 questions and the WHOQOL-Brief with 26 questions
Circadian rhythm | 12 months
  Munich Chronotype Questionnaire
Composite measure of Cognitive function | 12 months
  1) Mini Mental State Examination (MMSE); 2) Digit Span Test, 3) Verbal Fluency Test, 4) The Rey Auditory-Verbal Learning Test, 5) The Boston Naming Test, 6) Trail Making Test, 7) Stroop Color and Word Test, 8) Benton Visual Retention Test (is an assessment of visual perception, memory, and visuo-constructive abilities), 9) Beck Anxiety and Depression Inventory, 10) SYMPTOM CHECK LIST 90R- SCL90-R.
Ophthalmological assessment | 12 months
  Retinal and choroidal changes
Heart rate variability | 12 months
  Heart rate variability (HRV) The following HRV indices will be calculated in time and in frequency domains using 5-min segments as recommended by the European Society of Cardiology and North American Society of Pacing and Electrophysiology: the mean of all normal RR intervals (mean RR), the root mean square of successive differences of normal adjacent RR intervals (rMSSD), the low-frequency component (LF, 0.04 - 0.15 Hz) and the high-frequency component (HF, 0.15 - 0.5 Hz).
Cost-utility analysis measured by QALY | 60 months
  Quality adjusted years of life (QALY) obtained by the intervention will be calculated.
Change from Baseline Arterial Blood Pressure Monitoring (ABPM) at three months | 3 months
  24-h, diurnal, and sleep systolic and diastolic blood pressure. Systolic and diastolic dipping.
Change from Baseline Arterial Blood Pressure Monitoring (ABPM) at six months | 6 months
  24-h, diurnal, and sleep systolic and diastolic blood pressure. Systolic and diastolic dipping.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Martinez, MD, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (2):
- Brazil (2):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: Undecided